CLINICAL TRIAL: NCT03031756
Title: Efficacy of Glycine Powder Air-Polishing Combined With Scaling and Root Planing in the Treatment of Periodontitis and Halitosis: A Randomized Clinical Study
Brief Title: Efficacy of Glycine Powder Air-Polishing Combined With Scaling and Root Planing in the Treatment of Periodontitis and Halitosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Hasan Guney YILMAZ, Assoc Prof Dr, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 33-236-2015
Record Dates: First submitted 2017-01-16; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Halitosis
Keywords: Air polishing
MeSH Terms: conditions — Halitosis | interventions — Emergency Treatment; Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- test (Experimental): SRP was performed using routine ultrasonic (Piezon Master 700; EMS, Nyon, Switzerland) and hand instrumentation, glycine powder air-polishing (GPAP) was performed for 10 seconds per surface after the instrumentation (Air-Flows Perio Powder, EMS, Nyon, Switzerland) was applied using a Perio-Flows hand-piece connected to an airflow unit (Air-Flow Masters, EMS).
  Interventions: Device: glycine powder air-polishing (Air-Flows)Perio Powder; Device: ultrasonic (Piezon Master 700; EMS, Nyon, Switzerland)
- control (Active Comparator): In the control group, SRP was performed using routine ultrasonic (Piezon Master 700; EMS, Nyon, Switzerland) and hand instrumentation.
  Interventions: Device: ultrasonic (Piezon Master 700; EMS, Nyon, Switzerland)

INTERVENTIONS:
Device: glycine powder air-polishing (Air-Flows)Perio Powder
  Other Names: EMS, Nyon
  Arms: test
Device: ultrasonic (Piezon Master 700; EMS, Nyon, Switzerland)
  Other Names: EMS Piezon Master

SUMMARY:
The aim of this clinical study was to evaluate the clinical efficacy of using perio flow adjunctively with mechanical instrumentation on periodontal parameters and halitosis.

Sixty patients who presented with 4-6-mm probing pocket depth (PPD) were recruited for the study. Patients were randomly assigned to glycine powder air-polishing (GPAP) or control groups. For both groups PPDscores were recorded at the baseline and 1 month. Volatile sulphur compound (VSC) values were measured by a halimeter at the baseline, immediately after treatment, and at 7 days, 14 days and 1 month.

ELIGIBILITY:
Inclusion Criteria:

* In the present trial, patients who had at least three teeth with 4-6-mm periodontal pockets.

Exclusion Criteria:

* acute infectious oral lesions,
* furcation defects,
* using antibiotics for any reason in the last 4 weeks,
* periodontal treatment in the last 6 months and
* pregnant or lactating patients.

Ages: 28 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Periodontal Pocket Depth (PPD) | 30 day.
  PD were evaluated:at the follow-up sessions by the investigator with by marking a point on a 10 mm periodontal probe.

SECONDARY OUTCOMES:
halimeter values. | 30 day.
  The changes of Volatile Sulphure Compaunds by were evaluated with Halimeter Device at the follow-up sessions by the investigator. The Halimeter reads out in parts-per-billion (ppb) of volatile sulfur compounds.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Guney YILMAZ, DDS,PhD, Study Director — Near East University, Faculty of Dentistry

IPD SHARING:
Plan to Share IPD: No